CLINICAL TRIAL: NCT03669809
Title: Association Between Serum Metabolism Markers and Biological Rhythm
Brief Title: The Biological Rhythm of Human Metabolite
Status: Recruiting | Type: Observational
Sponsor: Shandong Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Jia-jun Zhao, Professor, Shandong Provincial Hospital
Other Study IDs: 20180326
Record Dates: First submitted 2018-04-03; First posted 2018-09-13 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2021-11

CONDITIONS: Rhythm Nodal; Metabolism and Nutrition Disorder; Metabolism Disorder, Lipid
Keywords: biological rhythm; metabolism; hormone; lipid; bile acids; obesity
MeSH Terms: conditions — Nutrition Disorders; Lipid Metabolism Disorders; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — serum，plasma, whole blood, urine, feces and seminal fluid
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- male, non-obese: male with BMI<28
- male, obese: male with BMI≥28
- female, non-obese: female with BMI<28
- female, obese: female with BMI≥28

SUMMARY:
The circadian regulation in mammals have been known for a long time. A special group of clock genes, organized in feedback loops, are responsible for the circadian regulation in both the SCN and peripheral organs. The central clock is mainly entrained by the light-dark cycle, while the peripheral ones in organs such as liver and intestine, are more influenced by the feeding-fasting cycles. The coordination of central and peripheral clocks is thought to be essential in the maintenance of physiological homeostasis.This study aim to investigate the association between biological rhythm and metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Male or female；
* Aged of 18 to 30 years old;

Exclusion Criteria:

* Presence of pituitary/hypothalamic disorders, polycystic ovarian syndrome， thyroid disorders, hypertension, malignant tumor, cardiac insufficiency，hepatic or renal insufficiency, gastrointestinal disorders and acute infection;
* Receiving psychotropic or hormonal medications including hormonal contraception and hormone therapies;
* Taking lipid-lowering agents or hypoglycemic agents and other drugs that known to influence cardiovascular health;
* Pregnancy or lactation women;
* Obviously poor compliance.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Adults aged of 18 to 30 years old.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2011-05-01; Primary Completion 2050-05-01 (Estimated); Study Completion 2050-05-01 (Estimated)

PRIMARY OUTCOMES:
circadian rhythms of serum lipid levels （the change of serum lipid levels within 24 hours） | Measured at baseline, and every 10 years during the 40-year follow-up period

SECONDARY OUTCOMES:
circadian rhythms of gonadal hormone and gonadotropin（the change of gonadal hormone and gonadotropin within 24 hours） | Measured at baseline, and every 10 years during the 40-year follow-up period
circadian rhythms of serum total bile acids（the change of serum total bile acids within 24 hours） | Measured at baseline, and every 10 years during the 40-year follow-up period
change in urine metabolite | Measured at baseline, and every 10 years during the 40-year follow-up period
change in intestinal flora | Measured at baseline, and every 10 years during the 40-year follow-up period
change in sperm quality | Measured at baseline, and every 10 years during the 40-year follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Jiajun Zhao, Study Chair — Shandong Provincial Hospital
Locations (1):
- Shandong Provincial Hospital, Jinan, Shandong, China